CLINICAL TRIAL: NCT00721825
Title: A Double-Blinded, Placebo-Controlled, Randomized Phase II Pilot Study to Investigate the Potential Efficacy of a Traditional Chinese Medicine NeuroAid In Enhancing Recovery After Stroke (TIERS)
Brief Title: Study of NeuroAid In Enhancing Recovery After Stroke
Acronym: TIERS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Moleac Pte Ltd. (Industry)
Responsible Party: Dr Kong Keng He - senior consultant, Tan Tock Seng Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Moleac
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2008-07

CONDITIONS: Stroke; Cerebral Infarction
Keywords: Stroke; Cerebral infarct; Rehabilitation; Double blind Randomized; Placebo controlled; Traditional Chinese Medicine; Neuroaid
MeSH Terms: conditions — Stroke; Cerebral Infarction | interventions — Neuroaid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Neuroaid
  Interventions: Drug: Neuroaid
- 2 (Placebo Comparator): Neuroaid matched placebo
  Interventions: Drug: Neuroaid matched Placebo

INTERVENTIONS:
Drug: Neuroaid — Neuroaid capsules, 4 capsules, three times per day, during one month
  Arms: 1
Drug: Neuroaid matched Placebo — Neuroaid matched placebo 4 capsules three times per day during one month
  Arms: 2

SUMMARY:
TIERS is a phase II to generate detailed preliminary data on the efficacy of NeuroAid in post-stroke recovery, and to assess the utility of the rehabilitation outcome measure instruments used.

ELIGIBILITY:
Inclusion Criteria:

* Subject had cerebral infarction confirmed by Computed Tomography (CT scan or Magnetic Resonance Imaging (MRI) imaging
* Presents within 1 month after stroke onset
* Presents with motor power of from grade 1 - 4/5 in at least one limb
* Has a pre-stroke modified Rankin score ≤ 1.
* Age between 21 and 80 years old
* Female subjects are eligible to participate in the trial if they are of non childbearing potential (hysterectomy or post-menopausal)
* Subject or legally acceptable representative is willing and able to provide written informed consent
* Subject and carer are willing and able to comply with investigational drug administration schedule.

Exclusion Criteria:

* Subject has received thrombolysis
* Subject has evidence of intra-cerebral hemorrhage on brain CT scan or MRI
* Subject has definite indication for full-dose or long-term anticoagulation therapy
* Subject has other significant non-ischemic brain lesion which could affect function disability
* Subject has co-existing systemic diseases: terminal cancer, renal failure (creatinine >200 μmol/L, if known), cirrhosis, severe dementia or psychosis
* Subject has a history of previous stroke/s
* Subject has participated in another clinical trial within the last three months
* Subject has aphasia or any other cognitive disabilities which prevent cooperation with study instructions
* Subject has dense hemiplegia (grade 0 motor power)
* Subject has haemoglobin level of <10mg/dl on admission
* Subject has a history of craniotomy or seizures

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer assessment | 4 weeks

SECONDARY OUTCOMES:
Functional Independence Measure (FIM) scale | 4 weeks and 8 weeks
Fugl-Meyer subscores | 4 weeks and 8 weeks
NIHSS and NIHSS subscores | 4 weeks and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Keng He Kong, MD, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Rehabilitation department, Singapore, Singapore